CLINICAL TRIAL: NCT03176550
Title: Effects of Somatosensory Electrical Simulation On Motor Function and Cortical Oscillations
Brief Title: Peripheral Stimulation Neural Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-123462
Record Dates: First submitted 2017-05-24; First posted 2017-06-05 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2020-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — TENS is performed using a commercially available device (ProStim, Alimed Inc, Dedham, Massachusetts, USA). One pair of 2 x 3.5 inches rectangular electrodes (Vermed ChroniCare TENS Electrodes, Vermed, Buffalo, NY, USA) are placed to simultaneously stimulate both median and ulnar nerves at the wrist, while a second pair of round 2 inch diameter electrodes are used to stimulate the radial nerve on the forearm. Bursts of electrical stimulation at 10 Hz (100 microsecond pulse width duration) are delivered to all nerves simultaneously for 2 hours.

SUMMARY:
Few patients recover full hand dexterity after an acquired brain injury such as stroke. Repetitive somatosensory electrical stimulation (SES) is a promising method to promote recovery of hand function. However, studies using SES have largely focused on gross motor function; it remains unclear if it can modulate distal hand functions such as finger individuation. The specific goal of this study was to monitor the effects of SES on individuation as well as on cortical oscillations measured using EEG, with the additional goal of identifying neurophysiological biomarkers.

DETAILED DESCRIPTION:
Participants with a history of acquired brain injury and distal upper limb motor impairments will receive a single two-hour session of SES using transcutaneous electrical nerve stimulation. Pre- and post-intervention assessments consist of the Action Research Arm Test (ARAT), finger fractionation, pinch force, and the modified Ashworth scale (MAS), along with resting-state EEG monitoring. We will assess for any association between SES and changes in motor outcome as measured using the ARAT, MAS and finger fractionation. In addition, EEG power analyses will be performed to determine if there are any differences between SES responders vs. non-responders.

ELIGIBILITY:
Inclusion Criteria:

* between 18-80 years old, with a history of an acquired brain injury resulting in residual hemiparesis or other motor deficits of the arm/hand equal to or more than 6 months prior to enrollment; and capacity to adhere with the schedule of interventions and evaluations determined in the protocol.

Exclusion Criteria:

* Subjects are excluded if they met any of the following criteria: currently pregnant; uncontrolled medical conditions; significant cognitive impairment on the Montreal Cognitive Assessment (MoCA ≤ 23); ≤ 10 degrees of active index finger range of motion; significant hand joint deformity; severe active alcohol or drug abuse; significant depression (PHQ-9 ≥15); baseline spasticity score (MAS) >3 for any joint tested (wrist and metacarpophalangeal joint flexion and extension); apraxia screen of Tulia (AST) <5; absent light touch, proprioception, pinprick and vibration sensation on the modified Nottingham Sensory Assessment; no upper limb strength against gravity; severe aphasia; or had an implanted pacemaker.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Action Research Arm Test (ARAT) | pre- and immediately post-stimulation
Change in Finger Fractionation | pre- and immediately post-stimulation

SECONDARY OUTCOMES:
Change in Modified Ashworth Scale (MAS) | pre- and immediately post-stimulation
Resting State EEG | pre- and immediately post-stimulation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tu-Chan AP, Natraj N, Godlove J, Abrams G, Ganguly K. Effects of somatosensory electrical stimulation on motor function and cortical oscillations. J Neuroeng Rehabil. 2017 Nov 13;14(1):113. doi: 10.1186/s12984-017-0323-1. PMID 29132379